CLINICAL TRIAL: NCT01211782
Title: A Phase 2-3, 6-12 Month, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Investigate the Effects of Daily Administration of AC-1204 in Subjects With Mild to Moderate Alzheimer's Disease Who Are APOE4(-)
Brief Title: AC-1204 Long-term Efficacy Response Trial (ALERT Protocol)
Acronym: ALERT
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study never started. Study was redesgined.
Sponsor: Cerecin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-10-006
Record Dates: First submitted 2010-09-24; First posted 2010-09-30 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; AD; AC-1204; ketogenic; ketosis
MeSH Terms: conditions — Alzheimer Disease; Ketosis | interventions — tricaprylin; Sunflower Oil; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AC-1204 (Experimental)
  Interventions: Drug: caprylic triglyceride
- Placebo (Placebo Comparator)
  Interventions: Drug: long-chain triglyceride

INTERVENTIONS:
Drug: caprylic triglyceride — oral, 20 gm, daily x 6 months
  Other Names: AC-1204
  Arms: AC-1204
Drug: long-chain triglyceride — oral, 14 gm, daily x 6 months
  Other Names: sunflower oil + maltodextrin
  Arms: Placebo

SUMMARY:
The study will evaluate the safety & efficacy of AC-1204, a ketogenic compound, administered orally on a daily basis for 6 months. Following the 6 month double-blind phase of the study, subjects may enroll in an optional 6 month open-label extension phase. Efficacy will be evaluated by standard tests of memory and cognition, along with other measurements of activities of daily living and quality of life. Safety will be assessed by frequency of adverse events and changes in laboratory test results. Subjects will be stratified and outcomes will be separately analyzed based on apolipoprotein E4 genotype (APOE4).

DETAILED DESCRIPTION:
Two primary outcome measures will be assessed in APOE4(-) patients:

1. differences from baseline between AC-1204 and placebo groups' ADAS-cog scores at 6 months
2. differences from baseline between AC-1204 and placebo groups' CIBIC+ scores at 6 months Secondary endpoints will include differences between AC-1204 & placebo groups' scores for these same instruments at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Males/females between age of 55 -85 years
* MMSE scores between 16-26
* Probable mild to moderate AD

Exclusion Criteria:

* Presence of other CNS disorders as alternative causes of dementia
* Type 1 or Type 2 diabetes
* Significant renal/hepatic disease

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Alzheimer's disease assessment scale - cognitive subscale (ADAS-cog) | 6 months
  change from baseline in ADAS-cog scores at 6 months in APOE4(-) patients

SECONDARY OUTCOMES:
Clinicians Interview Based Impression of Change with Caregiver Input (CIBIC+) | 6 months
  change from baseline in CIBIC+ scores at 6 months in APOE4(-) patients

CONTACTS AND LOCATIONS:
Overall Officials: Mildred Farmer, MD, Principal Investigator — Meridien Research
Locations (1):
- Meridien Research, St. Petersburg, Florida, United States